CLINICAL TRIAL: NCT03519061
Title: Impact of Budesonide Irrigations on Patients With Chronic Rhinosinusitis and Impact on Sinus Surgery Rates
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Unable to obtain FDA exemption
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Budesonide SInus Irrigations; 000001 (Other: Kaiser Permanente Southern California IRB)
Record Dates: First submitted 2018-04-26; First posted 2018-05-08 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Chronic Sinus Infection; Chronic Sinusitis; Chronic Sinusitis - Ethmoidal, Posterior; Chronic Sinus Congestion
MeSH Terms: interventions — Budesonide

STUDY DESIGN:
Intervention Model Description: Non randomized, single arm, prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): This is the group of enrollees who receive budesonide
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide — Nasal saline irrigations with budesonide

SUMMARY:
This study is intended to assess the impact of a 90 day course of high volume budesonide irrigations for patients who have failed other medical therapy and assessing the impact of the budesonide irrigations on the need for sinus surgery.

DETAILED DESCRIPTION:
Patient who meet eligibility requirements will be given the opportunity to use a budesonide saline rinse twice daily for 90 days. At the completion of this therapy, their clinical situation will be reassessed and patients will either proceed to surgery or not. If eligible patients choose not participate, they will be offered surgery up front. The study will be assessing symptom scores using the SNOT-22 validated patient reported symptoms score, CT scans, and other measures. The study hypothesizes that a significant portion of patients that otherwise would have progressed to surgery will no longer need to have surgery based upon improvements in their overall symptoms scores after using budesonise irrigations.

ELIGIBILITY:
Inclusion Criteria:

* adult (>18 yo)
* symptoms consistent with sinusitis for at least 12 weeks,
* undergone maximal medical therapy, including: extended course of antibiotics (21 days minimum), use of topical corticosteroids for a minimum of 6 weeks, use of saline rinses at least once a day for a minimum of 3 weeks
* CT showing evidence of chronic sinusitis.

Exclusion Criteria:

* pregnant women,
* age below 18,
* presence of nasal polyps or other nasal masses,
* failure to complete medical therapy,
* normal CT scan,
* intolerance to budesonide or saline irrigations via squeeze bottle (high volume, high flow).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-13 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
SinoNasal Outcome Test (SNOT 22) | 12 months
  Improvement in SNOT 22 scores, using a total score value. The total score can range from 0 to 110 in its composite score, with higher values indicating worse symptoms. The outcome would measure improvements beyond the Minimal Clinically Important Difference (MCID) score of 8.9 lower (lower indicating improvement of symptoms).

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanante Orange County, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No